CLINICAL TRIAL: NCT01722734
Title: Preserving ACTs - Text Reminders to Increase Adherence to ACT Treatment
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Günther Fink, Assistant Professor of International Health Economics, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19850-101
Record Dates: First submitted 2012-11-02; First posted 2012-11-07 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-02

CONDITIONS: Malaria
Keywords: Malaria; ACTs
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Patients in the control arm only got a generic health message at the end of the study.
- Short Message (Active Comparator): Patients in this arm receive six short text message reminders within 60 hours of treatment initiation at 12 hour intervals.
  Interventions: Behavioral: Text message reminders
- Long message (Active Comparator): Patients in this arm receive six long text message reminders (reminders including justification for why patients should finish medication) within 60 hours of treatment initiation at 12 hour intervals.
  Interventions: Behavioral: Text message reminders

INTERVENTIONS:
Behavioral: Text message reminders — Patients in the two treatment arms receive six short text message reminders within 60 hours of treatment initiation at 12 hour intervals to remind them to take their malaria medication as prescribed.
  Arms: Long message; Short Message

SUMMARY:
A randomized controlled trial was conducted to assess the effectiveness of text reminders sent to ACT users through an automated text messaging system short-message-system.

Study hypothesis: text message reminders increase adherence

DETAILED DESCRIPTION:
A randomized controlled trial was conducted to assess the effectiveness of text reminders sent to ACT users through an automated text messaging system short-message-system. Patients were enrolled at clinics and pharmacies upon receipt of ACTs and enrolled in the automated system for 3 days.

ELIGIBILITY:
Inclusion Criteria:

-subjects acquiring ACTs in Tamale, Ghana

Exclusion Criteria:

* subjects acquiring ACTs for non household members
* subjects under the age of 18
* subjects without access to cell phones
* subjects living more than 30 minutes from pickup location

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1140 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gunther Fink, PhD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Study site, Tamale, Northern Region, Ghana

REFERENCES:
- [Derived] Raifman JR, Lanthorn HE, Rokicki S, Fink G. The impact of text message reminders on adherence to antimalarial treatment in northern Ghana: a randomized trial. PLoS One. 2014 Oct 28;9(10):e109032. doi: 10.1371/journal.pone.0109032. eCollection 2014. PMID 25350546

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at all private and public facilities distributing Artemisinin-combination Therapies (ACTs).
Pre-assignment Details: Only subjects from the Tamale area with cell phones were included.
Groups:
- Control: Control group participants received only a message after five days informing them about the importance of using bed nets for malaria. No reminders to take ACTs were sent.
Period: Overall Study
Arm/Group | Control | Short Message | Long Message
Started | 554 | 277 | 309
Completed | 552 | 276 | 307
Not Completed | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Control: Patients in this group received only a generic malaria information message (use bed nets) at the end of the study.
- Total: Total of all reporting groups
Arm/Group | Control | Short Message | Long Message | Total
Number analyzed (Participants) | 554 | 277 | 309 | 1140
Age, Categorical [Count of Participants; unit: Participants] — Age is reported for the sick person in the household, which includes children in the care of adults, who were enrolled in the study and who received the message treatments.
  Participants
    <=18 years | 166 | 105 | 111 | 382
    Between 18 and 65 years | 342 | 158 | 166 | 666
    >=65 years | 46 | 14 | 32 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] — Age reflects age of the patient. For patients of age 18 and younger, caregivers were enrolled and interviewed and thus primary study subjects.
  years | 25.3 (17.7) | 23 (17.1) | 23.8 (17.8) | 24.3 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 302 | 152 | 180 | 634
  Male | 252 | 125 | 129 | 506
Region of Enrollment [Number; unit: participants]
  Ghana | 554 | 277 | 309 | 1140

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Adherence to Artemisinin-combination Therapy (ACT) Treatment
Description: Percentage of participants completing full ACT treatment regimen 70 hours after treatment initiation. Subjects were visited at home, and asked to report when each of the prescribed six doses were taken. Adherence was defined as the (self-reported) completion of all six doses.
Time Frame: 70 hours
Population: The number of subjects analyzed is smaller than the number of subjects enrolled due to missing data on adherence. A total of 30 observations were lost due to missing information on adherence - 16 in the control group, 9 in the short message group, and 5 in the long message group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Control: Subjects in this group received only one generic malaria message (use bed nets) at the end of the study.
Arm/Group | Control | Short Message | Long Message
Number analyzed (Participants) | 538 | 268 | 304
percentage of participants | 61.5 [57.39 to 65.648] | 69.0 [63.45 to 74.60] | 64.1 [58.72 to 69.56]

ADVERSE EVENTS:
Time Frame: Adverse effects were restricted to the 3 days monitoring period.
Groups:
- Control: Patients in this group received only a generic malaria message at the end of the study.
Arm/Group | Control | Short Message | Long Message
Serious Adverse Events (participants affected / at risk) | 0/554 | 0/277 | 0/309
Other Adverse Events (participants affected / at risk) | 0/554 | 0/277 | 0/309

LIMITATIONS AND CAVEATS:
Main outcome is self-reported adherence. Study was restricted to urban population with mobile phone ownership.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes